CLINICAL TRIAL: NCT02193542
Title: Prospective Observation Study of Incidence of Difficult Airway and Difficult Neuraxial Placement in Obstetric Patients
Brief Title: Incidence of Difficult Airway and Difficult Neuraxial Placement in Obstetric Patients
Acronym: DADB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Vice Chair, Faculty Development and Education; Director of Anesthesia, Center for Reproductive Medicine, Brigham and Women's Hospital
Other Study IDs: bwhobanes-DADB
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Indication for Care or Intervention Related to Labor or Delivery With Baby Delivered
Keywords: regional anesthesia; general anesthesia; obstetric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant patient: Pregnant woman presenting for vaginal or cesarean delivery

SUMMARY:
Anesthesiologists commonly administer pain relief during labor or providing anesthesia for cesarean delivery. Two main methods are used to achieve these goal: "Regional anesthesia" where the mother is given medication through a needle or catheter in her back and the mother is kept awake, or "General anesthesia", where the mother is given intravenous medication and is kept asleep.

Regional anesthesia uses a needle to enter a narrow space in the mother's back where medications can be given. In some patients, it takes longer to find this target space in the back. In emergency situation, however, there is often little time to find this space, and the backup method would be the general anesthesia technique.

If general anesthesia is required, a breathing tube needs to be inserted to help support the mother's breathing. In some patients, it is harder to insert the breathing tubes, so knowing this in advanced helps anesthesiologists create a safe plan for the patients. A lot of research has been done to determine factors that would predict which patients would need more time and preparation for general anesthesia and regional anesthesia.

The purpose of this study is to study how common it is for the pregnant patients who have a difficult regional and general anesthesia.

DETAILED DESCRIPTION:
Anesthesiologists commonly administer pain relief during labor or providing anesthesia for cesarean delivery. Two main methods are used to achieve these goal: "Regional anesthesia" where the mother is given medication through a needle or catheter in her back and the mother is kept awake, or "General anesthesia", where the mother is given intravenous medication and is kept asleep.

Regional anesthesia uses a needle to enter a narrow space in the mother's back where medications can be given. In some patients, it takes longer to find this target space in the back. In emergency situation, however, there is often little time to find this space, and the backup method would be the general anesthesia technique.

If general anesthesia is required, a breathing tube needs to be inserted to help support the mother's breathing. In some patients, it is harder to insert the breathing tubes, so knowing this in advanced helps anesthesiologists create a safe plan for the patients. A lot of research has been done to determine factors that would predict which patients would need more time and preparation for general anesthesia and regional anesthesia.

The purpose of this study is to study how common it is for the pregnant patients who have a difficult regional and general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman presenting for vaginal or cesarean delivery

Exclusion Criteria:

* Pregnant woman presenting for vaginal or cesarean delivery requiring urgent or emergent delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant woman presenting for vaginal or cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of difficult regional and general anesthesia | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Tsen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bucklin BA, Hawkins JL, Anderson JR, Ullrich FA. Obstetric anesthesia workforce survey: twenty-year update. Anesthesiology. 2005 Sep;103(3):645-53. doi: 10.1097/00000542-200509000-00030. No abstract available. PMID 16129992
- [Background] Hawkins JL. Anesthesia-related maternal mortality. Clin Obstet Gynecol. 2003 Sep;46(3):679-87. doi: 10.1097/00003081-200309000-00020. No abstract available. PMID 12972749
- [Background] Ross BK. ASA closed claims in obstetrics: lessons learned. Anesthesiol Clin North Am. 2003 Mar;21(1):183-97. doi: 10.1016/s0889-8537(02)00051-2. PMID 12698840
- [Background] Ellinas EH, Eastwood DC, Patel SN, Maitra-D'Cruze AM, Ebert TJ. The effect of obesity on neuraxial technique difficulty in pregnant patients: a prospective, observational study. Anesth Analg. 2009 Oct;109(4):1225-31. doi: 10.1213/ANE.0b013e3181b5a1d2. PMID 19762752
- [Background] Fettes PD, Jansson JR, Wildsmith JA. Failed spinal anaesthesia: mechanisms, management, and prevention. Br J Anaesth. 2009 Jun;102(6):739-48. doi: 10.1093/bja/aep096. Epub 2009 May 6. PMID 19420004